CLINICAL TRIAL: NCT00308685
Title: Chronic-Dose Safety and Efficacy Study of Albuterol-HFA-BAI (PROAIR™ HFA (Albuterol Sulfate) Breath Actuated Inhalation Aerosol) in Pediatric Asthmatics
Brief Title: Chronic-Dose Safety and Efficacy Study of Albuterol-HFA-BAI in Pediatric Asthmatics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IXR-303-25-167
Record Dates: First submitted 2006-03-28; First posted 2006-03-30 (Estimated); Results first posted 2022-02-24 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Asthma
Keywords: Asthma; Pediatric asthma
MeSH Terms: conditions — Asthma | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Albuterol-HFA-BAI (Experimental): ProAir(TM) HFA, Breath Actuated Inhalation Aerosol
  Interventions: Drug: Albuterol
- Placebo-HFA-BAI (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Albuterol — Albuterol 90mcg
  Arms: Albuterol-HFA-BAI
Drug: Placebo — Placebo
  Arms: Placebo-HFA-BAI

SUMMARY:
This study is designed to evaluate the repeat-dose safety and effectiveness of a bronchodilator inhaler relative to placebo (inactive drug inhaler) in children aged 4-11 years with asthma. The dosing period lasts three weeks and starts following a three-week run-in period.

ELIGIBILITY:
Inclusion Criteria:

* Persistent asthma of a minimum of six months duration that has been stable for at least four weeks prior to screening
* Male and female children aged 4-11 years, inclusive, with predicted forced expiratory volume in 1 second (FEV1) 60-90%
* Ability to perform spirometry
* Demonstrate 12% airways reversibility

Exclusion Criteria:

* Require continuous treatment with beta-blockers, monoamine oxidase inhibitors, tricyclic antidepressants, anticholinergics, and/or systemic corticosteroids
* Presence of any non-asthmatic clinically-significant acute or uncontrolled chronic diseases

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 95 (Actual)
Dates: Start 2006-06-10 (Actual); Primary Completion 2006-12-04 (Actual); Study Completion 2006-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, M.D., Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (14):
- United States (14):
  - Little Rock Allergy and Asthma, Little Rock, Arkansas
  - Allergy & Asthma Specialist Medical Group, Huntington Beach, California
  - Allergy & Asthma Associates of Santa Clara Valley Research Center, San Jose, California
  - William Storms Medical Research, Colorado Springs, Colorado
  - Colorado Allergy and Asthma Centers, PC, Denver, Colorado
  - Colorado Allergy and Asthma Centers, PC, Englewood, Colorado
  - Colorado Allergy and Asthma Centers, PC, Lakewood, Colorado
  - Southern Allergy & Asthma, PC, Savannah, Georgia
  - Sneeze, Wheeze & Itch Associates, Inc., Normal, Illinois
  - Clinical Research Institute, Minneapolis, Minnesota
  - The Asthma & Allergy Center, PC, Papillion, Nebraska
  - Allergy and Respiratory Center, Canton, Ohio
  - Allergy, Asthma & Clinical Research Center, Oklahoma City, Oklahoma
  - Pediatric Pulmonary Associates of North Texas, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Albuterol-HFA-BAI: Participants received albuterol
- Placebo-HFA-BAI: Participants received placebo
Period: Overall Study
Arm/Group | Albuterol-HFA-BAI | Placebo-HFA-BAI
Started | 50 | 45
Received at Least 1 Dose of Study Drug | 50 | 45
Completed | 47 | 40
Not Completed | 3 | 5
Not completed — Lost to Follow-up | 1 | 0
Not completed — Need to administer prohibited medication | 1 | 2
Not completed — Other than specified | 1 | 3

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Albuterol-HFA-BAI | Placebo-HFA-BAI | Total
Number analyzed (Participants) | 50 | 45 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.3 (2.22) | 8.8 (1.58) | 8.5 (1.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 26 | 53
  Male | 23 | 19 | 42
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 35 | 36 | 71
  Race: Black | 13 | 9 | 22
  Race: Asian | 1 | 0 | 1
  Race: Other | 1 | 0 | 1
Forced Expiratory Volume in 1 Second (FEV1) [Mean (Standard Deviation); unit: liters] — The baseline FEV1 was defined as the average of the 2 test-day (Day 22) predose (-0.5 and 0.0 hour prior to dosing) baseline FEV1 values.
  liters | 1.52 (0.44) | 1.61 (0.38) | 1.56 (0.42)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Percent Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) Observed up to 2 Hours Following Completion of Dosing (FEV1max%0-2) at Day 22
Description: The baseline FEV1 was defined as the average of the two predose measurements ( at -0.5 and 0.0 hour) on the test day (Day 22). The mean was obtained from the analysis of covariance (ANCOVA) adjusted for baseline FEV1 and the pooled investigational center.
Time Frame: Baseline (Predose at Day 22), 2 hours postdose at Day 22
Population: Intent-to-treat (ITT) population included all randomized participants who took at least 1 dose of the assigned study medication and had at least 1 postdose spirometry measurement.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Albuterol-HFA-BAI | Placebo-HFA-BAI
Number analyzed (Participants) | 50 | 45
percent change | 13.807 (0.954) | 8.644 (1.044)
Statistical Analysis 1: Comparison: Albuterol-HFA-BAI vs Placebo-HFA-BAI; Analysis was performed using an analysis of covariance (ANCOVA) with baseline FEV1 as covariate and fixed effects of pooled center and treatment group; Test type: Other; p = 0.0002, ANCOVA — Threshold for significance at 0.05 level; Difference in adjusted means = 5.163, 95% CI 2-sided [2.478 to 7.847]

2. Secondary Outcome: Baseline-Adjusted Area Under the Percent-Predicted FEV1 Versus Time Curve Over 6 Hours (PPFEV1 AUEC0-6) at Day 22
Description: Baseline-adjusted PPFEV1 AUEC0-6 on Study Day 22 was determined using both the Day 1 and Day 22 baselines.
Time Frame: Predose (30 and 5 minutes) and 15, 30, 45, 60, 120, 240, and 360 minutes postdose at Day 22
Population: ITT population included all randomized participants who took at least 1 dose of the assigned study medication and had at least 1 postdose spirometry measurement.
Measure: Mean (Standard Error); unit: percentage of predicted FEV1*hour
Arm/Group | Albuterol-HFA-BAI | Placebo-HFA-BAI
Number analyzed (Participants) | 50 | 45
percentage of predicted FEV1*hour
  PPFEV1 AUEC0-6 on Day 22 Using Day 22 Baseline | 29.473 (4.033) | 11.672 (4.476)
  PPFEV1 AUEC0-6 on Day 22 Using Day 1 Baseline | 43.182 (6.036) | 6.767 (6.572)

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 22
Description: Safety population included all randomized participants who received at least 1 dose of their assigned study medication.
Arm/Group | Albuterol-HFA-BAI | Placebo-HFA-BAI
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/45
Other Adverse Events (participants affected / at risk) | 0/50 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.